CLINICAL TRIAL: NCT04293744
Title: Acute Kidney Injury After Cardiac Surgery; A Prospective Randomized Study of Dextran Based and Crystalloid Priming Solutions (PRIMING II Trial)
Brief Title: Acute Kidney Injury After Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Priming II Trial
Record Dates: First submitted 2020-01-17; First posted 2020-03-03 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Surgical Procedures; Extracorporeal Circulation; Complications; Acute Kidney Injury
Keywords: Colloid priming solution; Cardiopulmonary bypass; Extracorporeal circulation; ECC; Acute Kidney Injury; AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colloid priming solution for ECC circuit (Experimental): Priming of ECC circuit with approximately 1200 mL PrimECC.
  Interventions: Device: Colloid priming solution for ECC circuit
- Standard priming solution for ECC circuit (Active Comparator): Priming of ECC circuit with approximately 1200 mL standard priming solution (crystalloid solution with or without mannitol addition as per routine of the participating clinic).
  Interventions: Device: Standard priming solution for ECC circuit

INTERVENTIONS:
Device: Colloid priming solution for ECC circuit — Prospective, multi-center, double-blinded, randomized, controlled clinical trial
  Arms: Colloid priming solution for ECC circuit
Device: Standard priming solution for ECC circuit — Prospective, multi-center, double-blinded, randomized, controlled clinical trial
  Arms: Standard priming solution for ECC circuit

SUMMARY:
PrimECC is a colloid priming solution for cardiopulmonary bypass/ extracorporeal circulation (ECC) based on Ringers Lactate, supplmeneted with Dextran 40 and Dextran 1. In a previous RCT comparing PrimECC with crystalloid priming fluid, patients in the PrimECC group experienced less hemolysis, less tubular cell injury and beneficial effect on the fluid balance. This study will investigate if, in a population at high risk of acute kidney injury (AKI), priming the ECC circuit with PrimECC instead of crystalloid solution will lead to a reduction of postoperative AKI. The hypothesis is that PrimECC, compared to crystalloid prime, will reduce postoperative AKI.

The study is a Swedish multicenter, double-blinded, randomized, controlled clinical trial. The trial will include 366 patients aged ≥18 years, scheduled for cardiac surgery with cardiopulmonary bypass, with an "Acute kidney injury risk score" ≥30% according to Birnie et al. (2014). The primary outcome of the study is the incidence of postoperative AKI of any stage according to the KDIGO creatinine criteria (serum-creatinine increase ≥ 27 μmol/l within 48 h or ≥ 50 % increase from baseline) within 96 hours after arrival to the ICU. Secondary outcomes are between-group differences in hemolysis, tubular cell injury (NAG-excretion), estimated GFR, and incidence of AKI of different stages according to the KDIGO creatinine criteria. In addition, differences in CNS (Tau, NFL, NSE, and S100B) and cardiac (TNT/TNI) injury markers will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Has signed and dated the EC approved informed consent
* Subject is ≥ 18 years of age
* Requires elective or urgent (non-emergency) cardiac procedure requiring the use of ECC.
* Preoperative "Acute kidney injury risk score" ≥30%, found at http://cardiacsurgeryleicester.com/our-research/acute-kidney-injury-risk-score-calculator/

Exclusion Criteria:

* Unable to give informed consent
* Known bleeding disorder
* Known intolerance or contraindication to dextran
* Acute Surgery (requires emergency cardiac procedure/surgery)
* Currently using an antithrombotic medication which has not been discontinued per institution protocol
* Malignancy; Surgery within 5 years or ongoing antitumoral treatment
* Has ongoing sepsis or endocarditis
* Requires pre-operative dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative AKI | Within 96 hours after ICU arrival
  Incidence of postoperative AKI of any stage according to the KDIGO creatinine criteria (serum-creatinine increase ≥ 27 μmol/l within 48 hours or ≥ 50 % increase from baseline)

SECONDARY OUTCOMES:
NAG excretion | 1 hour post initiation of ECC, at 1 hour after disconnection from ECC and 24 hours after disconnection from ECC.
  NAG-excretion (U-NAG/U-creatinine)
eGFR | Pre-operative and within 96 hours after ICU arrival
  pre-operative (day before surgery) compared to the highest post-operative value Measured value of pre-operative eGFR compared to the highest post-operative value within 96 hours after ICU arrival, calculated using the CKD-EPI formula
Incidence of AKI | Within 96 hours after ICU arrival
  Incidence of AKI of different stages according to the KDIGO creatinine criteria
Hemolysis | Pre-operative (after induction of anesthesia) and at 1 hour post initiation of ECC, 1 hour after disconnection from ECC and at 24 hours after disconnection from ECC.
  Hemolysis measured as free hemoglobin (PfHb)
CNS injury markers | Pre-operative (after induction of anesthesia), 1 hour after disconnection from ECC and at 24 hours after disconnection from ECC.
  Measured concentrations of CNS injury markers Tau, NFL, NSE, and S100B
Myocardial injury markers | Pre-operative (after induction of anesthesia) and at 1 hour after discontinuation of ECC and 24 hours after disconnection from ECC.
  Measured concentrations of myocardial injury markers TnI or TnT. TnI or TnT is chosen according to institutional standard

OTHER OUTCOMES:
Post-operative bleeding | The first 24 hours after disconnection from ECC
  Drain losses
Post-operative transfusions and use of hemostatic agents | The first 24 hours after disconnection from ECC
  Total transfusions and/or use of erythrocytes, plasma, thrombocytes, hemostatic pharmaceuticals

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Lannemyr, MD,PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Juvakka O, Wallinder A, Moller-Sorensen PH, Matschke K, Jeppsson A, Lannemyr L. Dextran vs. Crystalloid Priming Solution in Cardiac Surgery: A Randomized Trial on Acute Kidney Injury. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70139. doi: 10.1111/aas.70139. PMID 41144782